CLINICAL TRIAL: NCT04181853
Title: The Effect of Aerobic Exercise on Genetic Molecules Related With Metabolism
Brief Title: The Effect of Aerobic Exercise on Genetic Molecules
Acronym: xnx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, GULIN FINDIKOGLU, Associate Professor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 60116787-020/83243
Record Dates: First submitted 2019-11-23; First posted 2019-12-02 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Diabetes Mellitus, Type 2; Aerobic Exercise; Genetic Response
Keywords: Type 2 diabetes mellitus; exercise; aerobic
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The study has 3 arms
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants wil be making exercise. It is not possible to make participants blinded to the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High intensity interval exercise (Active Comparator): Participants with type 2 Diabetes mellitus in High intensity interval exercise (HIIE) group will make aerobic exercise using bicycle at high intensity followed by low intensity periods under observation in the hospital.
  Interventions: Other: exercise
- Moderate intensity continuous exercise (Active Comparator): Participants with type 2 Diabetes mellitus in Moderate intensity continuous exercise (MIC) group will make aerobic exercise using bicycle at moderate intensity during the session under observation in the hospital.
  Interventions: Other: exercise
- No Intervention: Control group (No Intervention): Participants with type 2 Diabetes mellitus in Moderate intensity continuous exercise (MIC) group will make aerobic exercise using bicycle at moderate intensity during the session under observation in the hospital.

INTERVENTIONS:
Other: exercise — aerobic exercise
  Arms: High intensity interval exercise; Moderate intensity continuous exercise

SUMMARY:
The aim of this study is to compare the effects of high intensity interval exercise and moderate intensity continuous exercise on some genetic molecules in patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Volunteers with type 2 diabetes mellitus will be evaluated in terms of any contra-indication that will restrain them from making exercise. 90 male or female volunteers who are suitable in terms of inclusion/exclusion criteria will be invited for the study. Volunteers will be randomly distributed to one of the 3 groups. Each group will contain 30 participants. 1. group will make aerobic exercise which is in the form of high intensity interval exercise 2.group will make aerobic exercise which is in the form of moderate intensity continuous exercise 3. Control group. Exercise groups will be cycling under observation in the hospital setting. Control group will make simple stretching exercises at home. Participants will be requested to complete a 3 months of exercise. They will be evaluated before and at the end of the 3 months of exercise with blood tests to measure genetic molecules related with metabolism.

ELIGIBILITY:
Inclusion Criteria:

Clinica diagnosis of type 2 Diabetes mellitus less than 10 years and more than 1 year.

* must have appropriate medical therapy and diet.
* must not be treated with insulin.
* must be exercising less than 210 minutes/ week

Exclusion Criteria:

* prominent cardiovascular disease
* coronary artery disease
* moderate to severe valvular disease
* atrial fibrillation
* untreated hypertension
* congenital heart disease
* retinopathy
* neuropathy
* macro albuminuria
* cerebrovascular disease
* ejection fraction less than 40
* body mass index greater than 35.
* prominent ischemic changes in EKG at rest or during exercise.
* cigarette or alcohol addiction
* on drugs that interferes with body fat distribution (such as insulin, thiazolidinediones

Ages: 30 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
genetic molecules | 12 weeks
  HbA1c level in the serum

CONTACTS AND LOCATIONS:
Overall Officials: Gulin Findikoglu, Assoc Prof, Principal Investigator — Pamukkale University,Medical Faculty, PMR Department
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No